CLINICAL TRIAL: NCT03393819
Title: Efficacy of Surgical Skin Preparation Solutions in Hip Arthroplasty Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lakehead University (Other)
Collaborators: Thunder Bay Regional Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Kurt Droll, Orthopaedic surgeon, Assistant Professor, Lakehead University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RP-002-01072013
Record Dates: First submitted 2018-01-03; First posted 2018-01-09 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Arthroplasty, Hip Replacement; Infection, Postoperative Wound
Keywords: antimicrobial skin solution; skin preparation
MeSH Terms: conditions — Surgical Wound Infection | interventions — DuraPrep; 2-Propanol; Chlorhexidine; Ethanol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinding of the participants and care providers after the assignment of the intervention is not possible as the two solutions are distinct, and one creates a unique discolouration of the skin. Those performing the laboratory analysis and reporting the results of the bacterial culture of will be blind to which treatment the participant was assigned (i.e. the label will not identify which group the participant belongs to).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Duraprep Surgical Solution (Experimental): Surgical site (hip) is prepared with Duraprep (iodine-alcohol) prior to surgery according to package instructions.
  Interventions: Drug: DuraPrep
- Chloraprep Surgical Solution (Experimental): Surgical site (hip) is prepared with Chloraprep (chlorhexidine-alcohol) prior to surgery according to package instructions.
  Interventions: Drug: ChloraPrep

INTERVENTIONS:
Drug: DuraPrep — DuraPrep surgical solution
  Other Names: Iodine Povacrylex and Isopropyl Alcohol
  Arms: Duraprep Surgical Solution
Drug: ChloraPrep — ChloraPrep surgical solution
  Other Names: chlorhexidine-alcohol
  Arms: Chloraprep Surgical Solution

SUMMARY:
This study will assess the efficacy of two of the most commonly used surgical skin-preparation solutions: Chloraprep (chlorhexidine-alcohol) and Duraprep (iodine-alcohol) at eliminating bacteria from the hip site by evaluating the residual bacteria present following surgical skin-preparation.

DETAILED DESCRIPTION:
Post-operative infections, although rare, can lead to significant patient morbidity and cost. A potential risk factor for the development of post-operative wound infection is the amount of bacterial skin flora present at the operative site at the time of surgery. Therefore, the use of an effective anti-microbial preoperative skin-preparation solution is essential in preventing the contamination of the surgical site and in turn the surgical wound.

Several different types of anti-microbial skin preparation solutions are presently used pre-operatively. However, there is currently no consensus on which solution is superior. Previous studies have investigated the efficacy of commonly used solutions in the shoulder, foot and spine, however the bacterial flora from these areas are likely different from the hip region. Thus the findings in the literature are not necessarily applicable to surgery involving the hip.

Because of the potentially devastating consequences of a surgical wound infection, ensuring effective skin preparation prior to surgery is critical. Therefore the identification of a superior skin-preparation solution for the elimination of bacterial pathogens, specific to the hip region, could potentially have considerable impact on the clinical care of patients undergoing hip arthroplasty surgery.

This study will assess the efficacy of two of the most commonly used surgical skin-preparation solutions: Chloraprep (chlorhexidine-alcohol) and Duraprep (iodine-alcohol), at eliminating bacteria from the hip site by evaluating the residual bacteria present following surgical skin-preparation.The primary outcome is as follows: positive culture rates of residual bacteria following surgical skin preparation. Secondary outcomes that will be evaluated is culture rates post-surgery (following skin closure) and acute (within 3 months) post-operative wound complications.

ELIGIBILITY:
Inclusion Criteria:

* Has consented for primary total hip arthroplasty by any of the following orthopaedic surgeons: Drs. Kurt Droll, Dave Puskas or Claude Cullinan
* Are capable of providing their own consent
* Are able to adequately communicate in English to undergo informed consent
* Has provided written, informed consent for the study

Exclusion Criteria:

* Previous hip arthroplasty
* Evidence of an open wound at the incision site
* Evidence of an abrasion in the vicinity of the planned incision
* Evidence of an active infection at or near the surgical site
* Evidence of an active infection elsewhere in the body
* Are chronically immunosuppressed e.g. transplant
* Is deemed not suitable for the study in the opinion of an investigator

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2014-10-29 (Actual); Primary Completion 2016-01-07 (Actual); Study Completion 2016-04-06 (Actual)

PRIMARY OUTCOMES:
Post-preparation skin swab | 4 minutes post-skin preparation
  bacterial culture rates following surgical skin preparation

SECONDARY OUTCOMES:
Post-operative skin swab | immediately after closure of the incision, before drape is removed from operative site
  bacterial culture rates following surgery
Post-operative wound complications | 3 months post-surgery
  wound complications at follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Droll, MD, Principal Investigator — TBRHSC

IPD SHARING:
Plan to Share IPD: No